CLINICAL TRIAL: NCT06047119
Title: Respiratory and Hemodynamic Targets During General Anesthesia - A Randomized Clinical Trial
Brief Title: Respiratory and Hemodynamic Targets During General Anesthesia
Acronym: GA-TARGETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lars Wiuff Andersen (Other)
Responsible Party: Sponsor-Investigator, Lars Wiuff Andersen, Associate Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 00005
Record Dates: First submitted 2023-08-10; First posted 2023-09-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Patients Undergoing General Anesthesia
MeSH Terms: interventions — Blood Pressure; Positive-Pressure Respiration; Tidal Volume

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Mean arterial blood pressure above 60 mmHg during general anesthesia and 2 hours after (Experimental)
  Interventions: Procedure: Blood pressure
- Mean arterial blood pressure above 70 mmHg during general anesthesia and 2 hours after (Experimental)
  Interventions: Procedure: Blood pressure
- Mean arterial blood pressure above 80 mmHg during general anesthesia and 2 hours after (Experimental)
  Interventions: Procedure: Blood pressure
- Systolic blood pressure above 90% of baseline during general anesthesia and 2 hours after (Experimental)
  Interventions: Procedure: Blood pressure
- Positive end expiratory pressure 5 cm H20 during general anesthesia (Experimental)
  Interventions: Procedure: Positive end expiratory pressure
- Positive end expiratory pressure 8 cm H20 during general anesthesia (Experimental)
  Interventions: Procedure: Positive end expiratory pressure
- Positive end expiratory pressure 10 cm H20 during general anesthesia (Experimental)
  Interventions: Procedure: Positive end expiratory pressure
- Tidal volume 5 ml/kg during general anesthesia (Experimental)
  Interventions: Procedure: Tidal volume
- Tidal volume 8 ml/kg during general anesthesia (Experimental)
  Interventions: Procedure: Tidal volume
- Tidal volume 10 ml/kg during general anesthesia (Experimental)
  Interventions: Procedure: Tidal volume
- Fraction of inspired oxygen 30% during general anesthesia and 2 hours after (Experimental)
  Interventions: Procedure: Fraction of inspired oxygen
- Fraction of inspired oxygen 80% during general anesthesia and 2 hours after (Experimental)
  Interventions: Procedure: Fraction of inspired oxygen

INTERVENTIONS:
Procedure: Blood pressure — Blood pressure targets during general anesthesia and 2 hours after
  Arms: Mean arterial blood pressure above 60 mmHg during general anesthesia and 2 hours after; Mean arterial blood pressure above 70 mmHg during general anesthesia and 2 hours after; Mean arterial blood pressure above 80 mmHg during general anesthesia and 2 hours after; Systolic blood pressure above 90% of baseline during general anesthesia and 2 hours after
Procedure: Positive end expiratory pressure — Positive end expiratory pressure during general anesthesia
  Arms: Positive end expiratory pressure 10 cm H20 during general anesthesia; Positive end expiratory pressure 5 cm H20 during general anesthesia; Positive end expiratory pressure 8 cm H20 during general anesthesia
Procedure: Tidal volume — Tidal volume during general anesthesia
  Arms: Tidal volume 10 ml/kg during general anesthesia; Tidal volume 5 ml/kg during general anesthesia; Tidal volume 8 ml/kg during general anesthesia
Procedure: Fraction of inspired oxygen — Fraction of inspired oxygen during general anesthesia and 2 hours after
  Arms: Fraction of inspired oxygen 30% during general anesthesia and 2 hours after; Fraction of inspired oxygen 80% during general anesthesia and 2 hours after

SUMMARY:
This trial is an investigator-initiated, multicenter, randomized, factorial, single-blind trial of multiple hemodynamic and respiratory targets during general anesthesia. These targets include blood pressure, positive end expiratory pressure, tidal volume, and fraction of inspired oxygen. Patients will be randomized to different targets using a factorial design, i.e., each patient is simultaneously randomized to four interventions. There will be five enrolling sites in the Central Denmark Region. 480 high-risk patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* American Society of Anesthesiologists (ASA) classification 3 to 5
* Planned endotracheal intubation with positive pressure ventilation
* Expected operating time ≥ 90 minutes
* Certain types of surgery

Exclusion Criteria:

* Inability to obtain consent (e.g., patient is unconscious, hyperacute surgery)
* Known or suspected pregnancy
* Out-patient/same-day surgery
* Intubated prior to surgery
* Clinical judgement by the anesthesiologist that any of the interventions could be potentially harmful to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Feasibility: Proportion of eligible patients randomized | Up to 90 days
  Eligible patients will be defined as those meeting all inclusion criteria and none of the exclusion criteria 1 to 4.
Feasibility: Proportion of patient with adherence to the assigned interventions | During surgery
  Adherence will be defined as follows:
  The allocated positive end expiratory pressure (± 1 cm H2O), tidal volume (± 1 ml/kg), and FiO2 (± 5%) is used in a minimum of 90% of the randomized patients for the duration of the surgery.
  Vasopressors/inotropes are only initiated and continued if the blood pressure declines below the allocated target in at least 60% of the patients and at least 60% of time during general anesthesia, i.e., 60% of the registered blood pressures should be within +/- 10 mmHg of the target when vasopressor/inotropes are administered.
Feasibility: Proportion of patients with separation of mean arterial pressure | During surgery
  We aim to achieve at least 5 mmHg separation in mean/median mean arterial pressure for the three blood pressure groups targeting mean arterial pressure.
Feasibility: Proportion of patients lost to follow-up | Up to 90 days
  We aim to obtain data from more than 90% of patients still alive at 30- and 90-days follow-up.

SECONDARY OUTCOMES:
Proportion of patients with pulmonary post-operative complications (composite) | 30 days
  A composite of the following based on European Perioperative Clinical Outcome definitions: Respirator infection, respirator failure, pleural effusion, atelectasis, pneumothorax, bronchospasms, and aspiration pneumonitis.
Proportion of patient with pneumonia | 30 days
  Based on the United States of America Centers for Disease Control and Prevention (CDC) definition of pneumonia
Proportion of patient with pulmonary embolism | 30 days
  Presence of pulmonary embolus on computerized tomography (CT) or magnetic resonance (MR) imaging, or a high probability of pulmonary embolus based on ventilation perfusion scan.
Proportion of patient with acute kidney injury | 30 days
  Composite of post-operative renal complications using Kidney Disease Improving Global Outcomes (KDIGO) criteria
Creatinine | 2 hours after the surgery
  Measured in umol/L
Creatinine | The day after the surgery
  Measured in umol/L
Proportion of patient with major adverse cardiac events | 30 days
  A composite of the following based on European Perioperative Clinical Outcome definitions: Non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure, new cardiac arrhythmia, and angina.
Troponin-I | 2 hours after the surgery
  Measured in ng/L
Troponin-I | The day after the surgery
  Measured in ng/L
Proportion of patients with myocardial injury after non-cardiac surgery | 3 days
  Post-operative troponin-I above the 99% percentile for the respective assay.
Alanine transaminase | 2 hours after the surgery
  Measured in U/L
Alanine transaminase | The day after the surgery
  Measured in U/L
Proportion of patients with emergence delirium | 2 hours after the surgery
  Based on the nursing delirium screening scale to evaluate emergence delirium 90-120 minutes after admission to the post-aesthesia care unit.
Proportion of patients with post-operative delirium | 7 days
  We will categorize delirium as delirium if this is either stated in the medical journal or retrospectively categorized as delirium if it meets pre-defined criteria based on the diagnostic and statistical manual of mental disorders, fifth edition from the American psychiatric association
Post-operative pain | 2 hours after the surgery
  Highest numeric rating scale (NRS) score (from 0 to 10 with higher scores indicating worse pain) documented
Opioid administered | 24 hours
  Total opioid administered using morphine equivalent units.
Proportion of patients with post-operative nausea and vomiting | 2 hours after the surgery
  Highest numeric rating scale (NRS) score (from 0 to 10 with higher scores indicating worse nausea and vomiting) documented
Antiemetic treatment | 24 hours
  Administered antiemetic treatment (ondansetron, dexamethasone, cyclizine, droperidol, metoclopramide) within the first 24 hours after the operation.
Proportion of patients with surgical site infections | 30 days
  Based on the United States of America Centers for Disease Control and Prevention (CDC) definition.
Clavien-Dindo grading of complications | 30 days
  In addition to reporting the individual post-operative complications, we will use the validated Clavien-Dindo classification to grade post-operative complications by the interventions needed.
Proportion of patients with intensive care unit admission | 30 days
  Both planned and unplanned stays at the intensive care unit.
Length of hospital stay | Up to 90 days
  Reported in days.
Days alive and out of the hospital | Within 30 days
  Reported in days. Patients that die during the 30 days, will receive a value of 0. All admissions at acute care hospitals in Denmark will be included in this outcome.
Proportion of patients with who die | 30 days
Proportion of patients with who die | 90 days
Health related quality of life | 30 days
  Based on the EQ-5D-5L questionnaire
Health related quality of life | 90 days
  Based on the EQ-5D-5L questionnaire
Proportion of patients with intraoperative complications | During surgery
  Specific complications occurring during the surgery: Bleeding, need of blood product transfusions, arrhythmia, pneumothorax, cardiac arrest, mortality.
Quality of recovery | 30 days
  Based on the quality of recovery-15 (QoR-15) score. The score ranges from 0-150 with higher scores indicating better recovery.
Quality of recovery | 90 days
  Based on the quality of recovery-15 (QoR-15) score. The score ranges from 0-150 with higher scores indicating better recovery.

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Gødstrup Regional Hospital, Gødstrup
  - Horsens Regional Hospital, Horsens
  - Randers Regional Hospital, Randers
  - Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
Six months after the publication of the last results, all de-identified individual patient data will be made available for data sharing. Procedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. Data will be completely anonymized according to Danish law.
  All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data. There will be no predetermined end date for the data sharing.
Supporting Information: Study Protocol
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered. Interested parties will be able to request the data by contacting the principal investigator. Authorship of publications emerging from the shared data will follow standard authorship guidelines from the International Committee of Medical Journal Editors and might or might not include authors from the steering committee depending on the nature of their involvement.

REFERENCES:
- [Background] Hoybye M, Lind PC, Holmberg MJ, Bolther M, Jessen MK, Vallentin MF, Hansen FB, Holst JM, Magnussen A, Hansen NS, Johannsen CM, Enevoldsen J, Jensen TH, Roessler LL, Klitholm MP, Eggertsen MA, Caap P, Boye C, Dabrowski KM, Vormfenne L, Henriksen J, Karlsson M, Balleby IR, Rasmussen MS, Paelestik K, Granfeldt A, Andersen LW. Fraction of inspired oxygen during general anesthesia for non-cardiac surgery: Systematic review and meta-analysis. Acta Anaesthesiol Scand. 2022 Sep;66(8):923-933. doi: 10.1111/aas.14102. Epub 2022 Jun 23. PMID 35675085
- [Background] Bolther M, Henriksen J, Holmberg MJ, Jessen MK, Vallentin MF, Hansen FB, Holst JM, Magnussen A, Hansen NS, Johannsen CM, Enevoldsen J, Jensen TH, Roessler LL, Caroe Lind P, Klitholm MP, Eggertsen MA, Caap P, Boye C, Dabrowski KM, Vormfenne L, Hoybye M, Karlsson M, Balleby IR, Rasmussen MS, Paelestik K, Granfeldt A, Andersen LW. Ventilation Strategies During General Anesthesia for Noncardiac Surgery: A Systematic Review and Meta-Analysis. Anesth Analg. 2022 Nov 1;135(5):971-985. doi: 10.1213/ANE.0000000000006106. Epub 2022 Oct 21. PMID 35703253
- [Background] Bolther M, Henriksen J, Holmberg MJ, Granfeldt A, Andersen LW. Blood pressure targets during general anaesthesia for noncardiac surgery: A systematic review of clinical trials. Eur J Anaesthesiol. 2022 Nov 1;39(11):903-905. doi: 10.1097/EJA.0000000000001703. Epub 2022 Jul 5. No abstract available. PMID 35797424
- [Background] Holst JM, Klitholm MP, Henriksen J, Vallentin MF, Jessen MK, Bolther M, Holmberg MJ, Hoybye M, Lind PC, Granfeldt A, Andersen LW. Intraoperative respiratory and hemodynamic strategies for reducing nausea, vomiting, and pain after surgery: Systematic review and meta-analysis. Acta Anaesthesiol Scand. 2022 Oct;66(9):1051-1060. doi: 10.1111/aas.14127. Epub 2022 Aug 22. PMID 35924389